CLINICAL TRIAL: NCT01223638
Title: The Prevalence of Hearing Loss Among Children With Congenital Hypothyroidism
Status: Withdrawn | Type: Observational
Why Stopped: written here by mistake
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dr. Yardena Tenenbaum - Rakover, HaEmek Medical Center, Israel
Other Study IDs: 0128-08-EMC
Record Dates: First submitted 2010-10-03; First posted 2010-10-19 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Congenital Hypothyroidism; Hearing Loss
Keywords: Congenital hypothyroidism(CH); Hearing loss among children with CH
MeSH Terms: conditions — Congenital Hypothyroidism; Hearing Loss | interventions — Hearing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Congenital hypothyroidism: Patient which were diagnosed with congenital hypothyroidism
  Interventions: Other: Audiometry
- Controls: Patients without any endocrine or hearing problems
  Interventions: Other: Audiometry

INTERVENTIONS:
Other: Audiometry — Audiometry

SUMMARY:
Congenital hypothyroidism (CH) occurs in 1:4000 live births. Neurological disturbances like speech delay, motor delay and lower IQ were reported in children with CH. Evidence from animal experiments indicate that CH is associated with high frequency of deafness. Morphological changes of the external and internal cholera hairs were reported in mutagenic mice with CH. Anatomical changes of the internal ear and low hearing threshold were reported in mice bearing Dual oxidase 2 (Duox2) gene mutations, which is responsible of oxidation of iodide. Knockout of Pax8 gene in mice resulted in both agenesis of thyroid gland and deafness. Early L-thyroxin therapy prevented the development of deafness in those mice. The expression of thyroid receptor α (TRα) in the external and internal cholera hairs in mice indicates that the thyroid hormones have an important role in the development of the internal ear.

The etiology of deafness in human is both genetic and environmental. The prevalence of deafness in live births is 1:1000 and among them 60% is genetic. Connexin 26 gene mutations are the most common cause of inherited deafness and account for about 40% of the genetic cases. In two conditions in human the coexistence of hypothyroidism and deafness were reported; Pendred syndrome and thyroid hormone resistance syndrome.

The prevalence of hearing loss in human with CH was explored in only few studies and the results are contrary.

The aim of the current study is to study the prevalence of hearing loss among children with CH and to compare the clinical, biochemical and genetic characteristics between subjects with hearing loss to those without hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients with congenital hypothyroidism aged 2-30 years

Exclusion Criteria:

* Hearing defects in the family
* Intrauterine infections
* Perinatal hypoxia
* Long term therapy with aminoglycosides
* Acoustic trauma in the past

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients aged 2-30 years with congenital hypothyroidism which are being followed at the Pediatric Endocrine Department at Ha'Emek Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Hearing Level | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ha'Emek Medical Center, Afula, Israel